CLINICAL TRIAL: NCT06481540
Title: Effect of the SpiroGym App on Voluntary Cough Strength in Parkinson's Disease
Brief Title: SpiroGym App-Aided Cough Rehabilitation
Acronym: ESApp PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Martin Srp, Ph.D., Ph.D., General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESApp PD
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease; Voluntary Peak Cough Strength; mHealth
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the experimental or the active control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the whole study protocol, patients did not receive information about testing the SpiroGym app. They will receive information that we are testing two types of expiratory muscle strength training programs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory muscle strength training + SpiroGym application (Experimental): The experimental arm will undergo 8 weeks of expiratory muscle strength training coupled with SpiroGym app.
  Interventions: Device: Expiratory muscle strength training + SpiroGym application
- Expiratory muscle strength training (Active Comparator): The experimental arm will undergo 8 weeks of expiratory muscle strength training.
  Interventions: Device: Expiratory muscle strength training

INTERVENTIONS:
Device: Expiratory muscle strength training + SpiroGym application — Participants will performe an intensive home-based expiratory muscle training programme using an Expiratory Muscle Trainer (EMST150; Aspire Products, LLC, United States), which provide a pressure- threshold range from 30 to 150 cmH20. EMST therapy sessions will be completed at home on 5 days of the patients choosing per week. Participants will be instructed to perform five sets of five forceful expirations coupled with SpiroGym app. per training session for 8 weeks (intensive training period). After this period, participants will perform an additional 16 weeks of maintenance EMST. EMST therapy sessions will be completed at home on two days (minimum) of the participant's choosing each week.
  Arms: Expiratory muscle strength training + SpiroGym application
Device: Expiratory muscle strength training — Participants will performe an intensive home-based expiratory muscle training programme using an Expiratory Muscle Trainer (EMST150; Aspire Products, LLC, United States), which provide a pressure- threshold range from 30 to 150 cmH20. EMST therapy sessions will be completed at home on 5 days of the patients choosing per week. Participants will be instructed to perform five sets of five forceful expirations per training session for 8 weeks (intensive training period).After this period, participants will perform an additional 16 weeks of maintenance EMST. EMST therapy sessions will be completed at home on two days (minimum) of the participant's choosing each week.
  Arms: Expiratory muscle strength training

SUMMARY:
The pilot study by Srp et al. (2021) proved that the SpiroGym app was feasible for supporting expiratory muscle strength training (EMST) in Parkinson's disease (PD) patients. Two weeks of intensive EMST coupled with SpiroGym were sufficient to significantly improve the participants' voluntary peak cough flow (PCF). The improvement was quantitatively comparable to the results of other intensive EMST studies with longer durations. When interpreting such rapid improvement, the impact of SpiroGym's visual feedback was considered. It was assumed that visual feedback increased training effort compared to regular training without immediate control. However, comparative studies were required to verify the possible additional effects of visual feedback on voluntary PCF compared to EMST without feedback.

DETAILED DESCRIPTION:
Goal: To explore the visual feedback effect of the SpiroGym app in EMST on voluntary peak cough

Hypothesis 1: Change in voluntary peak cough flow will be higher in the experimental group than in the active control group after 8weeks and 24 weeks of EMST.

Study Design: A double-blind, randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinsons disease
* Stable dopaminergic medication (stable dose for at least 1 month)

Exclusion Criteria:

* Other neurological disorders
* Difficulty complying due to neuropsychological dysfunction (dementia with a score of less - - than 19 on the Montreal Cognitive Assessment)
* Breathing disorders or diseases
* Smoking in the past 5 years
* Uncontrolled hypertension

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Voluntary peak cough flow | 1 week before baseline, baseline, 8 weeks, 24 weeks
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srp M, Korteova R, Kliment R, Jech R, Ruzicka E, Hoskovcova M. Expiratory Muscle Strength Training in Patients with Parkinson's Disease: A Pilot Study of Mobile Monitoring Application. Mov Disord Clin Pract. 2021 Aug 4;8(7):1148-1149. doi: 10.1002/mdc3.13313. eCollection 2021 Oct. No abstract available. PMID 34631956
- [Background] Troche MS, Curtis JA, Sevitz JS, Dakin AE, Perry SE, Borders JC, Grande AA, Mou Y, Vanegas-Arroyave N, Hegland KW. Rehabilitating Cough Dysfunction in Parkinson's Disease: A Randomized Controlled Trial. Mov Disord. 2023 Feb;38(2):201-211. doi: 10.1002/mds.29268. Epub 2022 Nov 7. PMID 36345090
- [Background] Troche MS, Rosenbek JC, Okun MS, Sapienza CM. Detraining outcomes with expiratory muscle strength training in Parkinson disease. J Rehabil Res Dev. 2014;51(2):305-10. doi: 10.1682/JRRD.2013.05.0101. PMID 24933728
- [Background] Reyes A, Castillo A, Castillo J. Effects of Expiratory Muscle Training and Air Stacking on Peak Cough Flow in Individuals with Parkinson's Disease. Lung. 2020 Feb;198(1):207-211. doi: 10.1007/s00408-019-00291-8. Epub 2019 Nov 12. PMID 31720808